CLINICAL TRIAL: NCT05347680
Title: A Prospective and Randomized Study Comparing Fiberoptic Intubation Through the New Intubating Laryngeal Tube Suction and the Ambu AuraGain in Adult Patients Secondary IDs:
Brief Title: A Comparison Between the Intubating Laryngeal Tube Suction and the Ambu AuraGain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0132-16
Record Dates: First submitted 2022-04-03; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Difficult Intubation
Keywords: fiberoptic; supraglottic; Laryngeal Tube; intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intubating laryngeal Tube Suction (Active Comparator): Fiberoptic Intubation through intubating laryngeal Tube Suction
  Interventions: Device: Intubating Laryngeal Tube Suction
- Ambu AuraGain Laryngeal Mask (Active Comparator): Fiberoptic Intubation through Ambu AuraGain Laryngeal Mask
  Interventions: Device: Ambu AuraGain Laryngeal Mask

INTERVENTIONS:
Device: Intubating Laryngeal Tube Suction — Intubating Laryngeal Tube Suction
  Arms: intubating laryngeal Tube Suction
Device: Ambu AuraGain Laryngeal Mask — Ambu AuraGain Laryngeal Mask
  Arms: Ambu AuraGain Laryngeal Mask

SUMMARY:
The intubating Laryngeal Tube Suction-Disposable is a new version of the Laryngeal Tube-Suction. It has a ventilator channel with a 13.5mm internal diameter, which enables the passage of an Endotracheal Tube with fiberoptic guidance. This study was designed to assess the Time fiberoptic endotracheal intubation using iLTS-D, in comparison with the and Ambu® AuraGain™ in adult patients.

DETAILED DESCRIPTION:
The intubating Laryngeal Tube Suction-Disposable is a new version of the Laryngeal Tube-Suction. It has a ventilator channel with a 13.5mm internal diameter, which enables the passage of an Endotracheal Tube with fiberoptic guidance. This study was designed to assess the Time of fiberoptic endotracheal intubation using iLTS-D, in comparison with the and Ambu® AuraGain™ in adult patients.

Detailed Description: The intubating Laryngeal Tube Suction-Disposable (iLTS-D) (VBM Medizintechnik GmbH, Sulz, Germany) is a new updated version of the Laryngeal Tube-Suction Disposable (LTS-D) It has a ventilator channel with a 13.5mm internal diameter, which enables the passage of an Endotracheal Tube (ETT) with fiberoptic guidance. Similarly as in to the LTS-D, the iLTS-D also has a separate channel for the purpose of placement of gastric tubes placement up to a size of 18 Fr.

The iLTS-D comes in one size. According to the depth of insertion, this device is equivalent to size 4 for patients height 175 to 190 cm tall, or size 5 for patients taller than 190 cm. The iLTS-D is provided by the manufacturer with a compatible 7.5 mm ETT and with a plastic stabilizer for removal of the device.

The current randomized study was designed to assess the success rate fiberoptic endotracheal intubation using iLTS-D, in comparison with the and Ambu® AuraGain™ in adult patients under general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiology I and II

Exclusion Criteria:

* Difficult intubation
* Cervical pathology
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Time to perform fiberoptic intubation through supraglottic device in second | 120 seconds
  Time to perform endotracheal fiberoptic intubation through supraglottic device in second

SECONDARY OUTCOMES:
Success to obtain fiberoptic intubation through supraglottic device in second | 120 seconds
  Success to obtain endotracheal fiberoptic intubation through supraglottic device in second

CONTACTS AND LOCATIONS:
Overall Officials: Luis Gaitini, Prof, Principal Investigator — Bani Zion Medical Center Haifa ISRAEL
Locations (1):
- Luis A Gaitini M.D., Haifa, Israel

IPD SHARING:
Plan to Share IPD: No